CLINICAL TRIAL: NCT02875704
Title: Oxidative Stress In Stargardt Disease, Age Related Macular Degeneration and Diabetic Retinopathy
Status: Terminated | Type: Observational
Why Stopped: There was no significant difference in our outcome measures between patients with disease versus controls suggesting that our hypothesis is not substantiated. Since this was the major objective of the study we decided to terminate the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00112564; OXI-SAD (Other: Other)
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2022-06

CONDITIONS: Stargardt Disease; Diabetic Retinopathy; Macular Degeneration (Age Related)
Keywords: DR; AMD
MeSH Terms: conditions — Stargardt Disease; Diabetic Retinopathy; Macular Degeneration | interventions — Paracentesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will only be used for measurement of biomarkers of oxidative stress
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stargardt disease, AMD, DR patients: Stargardt disease, Age Related Macular Degeneration, Diabetic Retinopathy patients
  Interventions: Other: Anterior Chamber (AC) Tap
- Controls: Patients without retinal disease who will be undergoing cataract surgery
  Interventions: Other: Anterior Chamber (AC) Tap

INTERVENTIONS:
Other: Anterior Chamber (AC) Tap — Aqueous Samples will be collected for measurement of biomarkers
  Other Names: AC Tap

SUMMARY:
In this study, markers of oxidative stress will be measured in the aqueous humour of stargardt disease, age related macular degeneration and diabetic retinopathy patients compared to controls.

DETAILED DESCRIPTION:
People with Stargardt disease, age related macular degeneration (AMD) and diabetic retinopathy (DR) have decrease in central vision from damage to photoreceptors. One of the mechanisms causing damage is high levels of oxygen in the eye. This damage produces specific biomarkers that can be measured in eye fluid (aqueous humor). In this study, these biomarkers will be assessed in people with Stargardt disease, age related macular degeneration and diabetic retinopathy, compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age at least 18 years
* For the study group, patients diagnosed with Stargardt disease, age related macular degeneration and diabetic retinopathy by the investigators, based on clinical phenotype
* For the control group, patients with no retinal disease undergoing cataract surgery will be eligible.

Exclusion Criteria:

• None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stargardt disease, AMD, DR patients and controls
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Aqueous levels of oxidized adducts on protein (i.e. oxidative biomarker) in patients with stargardt disease, AMD, DR and controls | Baseline
  Baseline = Day of clinic visit for stargardt disease, AMD, DR patients and day of surgery for patients undergoing cataract surgery. No follow up is required.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No